CLINICAL TRIAL: NCT02311322
Title: Genetic Causes of Growth Disorders
Status: Terminated | Type: Observational
Why Stopped: PI left NIH
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150022; 15-CH-0022
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Short Stature; Growth Disorder; Syndromic Growth Disorder; Tall Stature
Keywords: Growth Disorder; Growth; Exome Sequencing
MeSH Terms: conditions — Dwarfism; Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, saliva, DNA extracted from whole blood or saliva, plasma, serum, urine, skin biopsy, hair follicles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with growth disorders: Children with growth disorders
- Family members of subjects with growth disorders: Family members of subjects with growth disorders

SUMMARY:
Background:

- Some growth disorders are caused by a change in genes. Genes are the instructions the body uses to function. Changes in genes often cause them not to work correctly. Researchers want to use a new technology called exome sequencing, to look at many genes at once. This is done by looking at DNA from blood or saliva in a lab. This method may help find the cause of disorders that researchers haven t been able to find using past methods.

Objectives:

- To better understand genetic causes of growth disorders.

Eligibility:

- Children and adults with growth disorders and their family members.

Design:

* Participants will give a small sample of blood and/or saliva.
* Researchers will purify DNA from the sample. They will perform exome sequencing and other tests to look for changes in genes. Some participants may receive limited or no genetic tests. Researchers will let them know if exome sequencing is performed.
* Participants may have a medical history, physical exam, and lab tests. They may have x-rays or ultrasound tests to study the disorder in their family.
* Some participants may be recommended for a specific genetic test from a commercial lab. They may have to pay for that test.
* Participants will be told about test results that relate to the growth disorder. This may happen up to years after the testing. They may have to give another blood and/or saliva sample.
* Some participants may get results about other health conditions. This will only happen if the information would help the person or their family protect their health. They may have to give another blood and/or saliva sample.

DETAILED DESCRIPTION:
Children often present to pediatricians and pediatric endocrinologists because of abnormal body growth, including both childhood growth failure and, less commonly, overgrowth. Sometimes the cause is evident, for example, growth hormone deficiency for growth failure and growth hormone excess for overgrowth. In other children, the etiology remains unknown despite extensive evaluation, resulting in the unhelpful diagnosis of severe idiopathic short stature or tall stature. These conditions are quite heterogeneous, including children with isolated growth disorders and others who also have other abnormalities such as developmental delay or a constellation of congenital anomalies (syndromic growth disorders). Some cases of severe growth disorders have a polygenic inheritance while others appear to be inherited as a monogenic trait - recessive, dominant or X-linked. Because of recent advances in DNA sequencing technology, it is now feasible to sequence the exome (portion of the genome that encodes gene exons) in families with monogenic disorders and thereby determine the underlying molecular etiology.

We therefore propose a study to identify novel genetic causes of idiopathic growth disorders using whole-exome sequencing. The primary goal of this study is to identify novel causes of childhood growth disorders in order to improve clinical diagnosis, to provide a more precise characterization of associated medical problems, prognosis, and response to treatment based on etiology, and to gain new insights into the regulation of human growth, which may eventually lead to new therapeutic approaches.

Subjects will include children and adults with a clearly recognizable phenotype that includes either short stature or tall stature and a pedigree that strongly suggests a monogenic inheritance. Both syndromic and non-syndromic growth disorders and both proportionate and disproportionate growth disorders will be included. Affected and unaffected family members (who have informative meiotic inheritance relationships to the proband or index case) will also be studied because of their importance for this genetic approach. The phenotype will be characterized by medical history, physical exam, body measurements, and laboratory evaluation. Blood and saliva samples will be collected for whole-exome sequencing and single nucleotide polymorphism (SNP) array analysis. Candidate sequence variants will typically be verified by Sanger sequencing.

ELIGIBILITY:
* INCLUSION CRITERIA:

If a subject meets any one of these criteria, he/she will potentially be eligible to participate:

* Short stature (height less than - 2 SDS), either currently or previously - or
* Tall stature (height greater than + 2 SDS) or
* Bone age delay (greater than 3 years) or
* Bone age advancement (>1.5 years) or
* Predicted adult height < - 2SD
* Predicted adult height - mid-parental height < -2SDS or > 2SDS
* Growth disorder that was treated promptly, thus maintaining the child s height within the normal range, e.g. a subject with congenital growth hormone deficiency or multiple pituitary hormone deficiency of unknown genetic etiology who received growth hormone treatment beginning in early life or
* Family member of subjects who meet any of the above criteria
* Subjects have a current height at a low normal percentile but has short adult height prediction based on bone age (> 5 inches shorter than mid-parent height)
* Any subject who has more than one of the above criteria and elevated DHEA-S concentration for age

In addition, subjects are only eligible, if, the pedigree suggests a monogenic inheritance, and, in the judgement of the investigators, there is a reasonable likelihood of identifying a novel gene responsible for the condition.

Investigators may recruit study subjects through The Genomic Ascertainment Cohort (TGAC) to identify specific subjects with sequence variants in genes of interest associated with growth disorders to investigate the phenotype spectrum, regardless of the above criteria.

Investigators may recruit study additional subjects through the NIDDK repository to identify specific subjects with sequence variants in genes of interest associated with growth disorders to investigate the phenotype spectrum, regardless of the above criteria. Investigators may first identify subjects with height < 3rd% from these cohorts, request their DNA samples and sequence their DNA to identify a variant in a gene of interest.

If subjects have abnormal bone age x-ray findings, investigators may use the findings as a maker for chondrodysplasia and study subjects with the findings. To recruit subjects, bone age x-rays obtained under teaching protocol (00-CH-0180 and 16-CH-0113) may be reviewed. If the subjects with abnormal findings are still followed by NIH, this study will be introduced to the patient and family. However, if subjects had been discharged from NIH care, they will not be re-contacted but their data may be still included in the prevalence of the abnormal finding. If collaborators wish to review their bone age x-rays obtained from their patients with short stature to identify the eligible subjects, they will obtain approval from their IRB. If some subjects are identified and the family agrees to participate, then collaborators refer them to our research team.

EXCLUSION CRITERIA:

* A non-genetic disorder or condition, either congenital or acquired, that explains the growth abnormality, for example, pituitary injury, chronic thyroiditis, whole body irradiation, or celiac disease.
* In the opinion of the investigators, there is an established diagnosis of a genetic disorder or condition that explains the growth abnormality and for which the molecular genetic etiology has already been identified, for example, SHOX deficiency, hypochondroplasia, or Noonan syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects with growth disorders
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
SNP array and whole exome sequencing data | 1-5 years
  identification of the causal variant

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Jee, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jee YH, Gangat M, Yeliosof O, Temnycky AG, Vanapruks S, Whalen P, Gourgari E, Bleach C, Yu CH, Marshall I, Yanovski JA, Link K, Ten S, Baron J, Radovick S. Evidence That the Etiology of Congenital Hypopituitarism Has a Major Genetic Component but Is Infrequently Monogenic. Front Genet. 2021 Aug 11;12:697549. doi: 10.3389/fgene.2021.697549. eCollection 2021. PMID 34456972
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-CH-0022.html